CLINICAL TRIAL: NCT00453648
Title: Efficacy of Daily Consumption of Sweet Potatoes for Increasing Total Body Vitamin A Pool Size, and the Effect of Consumption of Sweet Potatoes on Iron and Zinc Absorption in Bangladeshi Women of Reproductive Age
Brief Title: Impact of Consumption of Orange-fleshed Sweet Potatoes on the Vitamin A Status of Bangladeshi Women of Reproductive Age
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 200513770; Harvest Plus 8027 (Other Grant/Funding Number: Harvest Plus Program); Harvest Plus 8033 (Other Grant/Funding Number: Harvest Plus Program)
Record Dates: First submitted 2007-03-27; First posted 2007-03-29 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Vitamin A Deficiency
Keywords: stable isotopes; vitamin A; beta-carotene; orange-fleshed sweet potatoes; iron; zinc; absorption; bioavailability; vitamin A equivalency; Bangladesh; women
MeSH Terms: conditions — Vitamin A Deficiency

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- White-fleshed Sweet Potato (Placebo Comparator): 0 ug retinol activity equivalents (RAE)/d as boiled white-fleshed sweet potatoes (WFSP) and a corn oil capsule, 6d/wk for 10 wk
  Interventions: Other: White-fleshed sweet potatoes
- Orange-fleshed Sweet Potato (boiled) (Experimental): 600 ug RAE/d as boiled orange-fleshed sweet potato and a corn oil capsule, 6d/wk for 10 wk
  Interventions: Other: Orange-fleshed sweet potatoes (boiled)
- Orange-fleshed Sweet Potato (fried) (Experimental): 600 ug RAE/d as fried orange-fleshed sweet potato and a corn oil capsule, 6d/wk for 10 wk
  Interventions: Other: Orange-fleshed sweet potatoes (fried)
- White-fleshed Sweet Potato and retinyl palmitate capsule (Active Comparator): 0 ug RAE/d as white-fleshed sweet potato and 600 ug retinol/d as retinyl palmitate, 6d/wk for 10 wk
  Interventions: Other: WFSP and capsule of retinyl palmitate

INTERVENTIONS:
Other: White-fleshed sweet potatoes
  Arms: White-fleshed Sweet Potato
Other: Orange-fleshed sweet potatoes (boiled)
  Arms: Orange-fleshed Sweet Potato (boiled)
Other: Orange-fleshed sweet potatoes (fried)
  Arms: Orange-fleshed Sweet Potato (fried)
Other: WFSP and capsule of retinyl palmitate
  Arms: White-fleshed Sweet Potato and retinyl palmitate capsule

SUMMARY:
The primary purpose of this study is to determine whether daily consumption of orange-fleshed sweet potatoes increases the vitamin A status of Bangladeshi women of reproductive age. Secondary purposes of the study are to determine whether consumption of orange-fleshed sweet potatoes has an effect on the intestinal absorption of dietary iron or dietary zinc in Bangladeshi women of reproductive age.

DETAILED DESCRIPTION:
Biofortification of plant source foods is a promising strategy for increasing dietary vitamin A intake and vitamin A status in populations at risk of deficiency. The primary purposes of this study are:

1. to assess the efficacy of daily consumption of boiled or fried orange-fleshed sweet potatoes (OFSP) for increasing the vitamin A status of non-pregnant, non-lactating Bangladeshi women, and
2. to estimate the relative vitamin A equivalency of beta-carotene from the two different preparations of OFSP (boiled or fried).

Secondary purposes are to assess the effect of daily consumption of OFSP on intestinal absorption of iron and zinc. Specifically, 120 non-pregnant, non-lactating women at risk of vitamin A deficiency will be randomly assigned to one of the following 4 treatment groups to receive, 600 micrograms RAE/d, 6 d/wk, for 60 days as either:

1. boiled OFSP
2. fried OFSP
3. retinyl palmitate, or 0 micrograms RAE/d as white-fleshed sweet potato (WFSP)

The paired stable isotope dilution technique will be used to estimate total body vitamin A pool size before and after 60-days of supplementation. The efficacy of consumption of OFSP will be assessed by comparing the mean change in vitamin A pool size in the OFSP groups to the mean change in vitamin A pool size in the negative control group (WFSP group). Relative vitamin A equivalency factors will be estimated by comparing the mean change in vitamin A pool size in the OFSP groups with the mean change in vitamin A pool size in the retinyl palmitate group. Intestinal iron absorption and iron status will be assessed before and after the 60-day supplementation period in a subset of women (n=50); and intestinal zinc absorption and zinc status will be assessed after the 60-day supplementation period (n=50). Intestinal absorption of iron and zinc will be compared by treatment group to determine whether consumption of OFSP has any effect on iron or zinc absorption in these women.

ELIGIBILITY:
Inclusion Criteria:

* Serum retinol concentration < 1.12 umol/L
* Serum C-reactive protein concentration < 10 mg/L

Exclusion Criteria:

* Pregnant
* Lactating
* Diarrhea within past week
* Severe anemia (< 9g Hb/dL)
* Symptoms of nightblindness
* Clinical symptoms of xerophthalmia
* Chronic disease

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 130 (Actual)
Dates: Start 2006-03; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Total body vitamin A pool size | 3 years

SECONDARY OUTCOMES:
Iron absorption | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Marjorie J Haskell, PhD, Principal Investigator — University of California, Davis; Kenneth H Brown, MD, Principal Investigator — University of California, Davis; Kazi Jamil, MBBS, PhD, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh

REFERENCES:
- [Derived] Jamil KM, Brown KH, Jamil M, Peerson JM, Keenan AH, Newman JW, Haskell MJ. Daily consumption of orange-fleshed sweet potato for 60 days increased plasma beta-carotene concentration but did not increase total body vitamin A pool size in Bangladeshi women. J Nutr. 2012 Oct;142(10):1896-902. doi: 10.3945/jn.112.164830. Epub 2012 Aug 29. PMID 22933750